CLINICAL TRIAL: NCT02772315
Title: Performance of an Omics-signature in the Diagnosis and Prognosis of Endocrine and Primary Hypertension
Brief Title: Omics Signature in the Diagnosis of Hypertension
Acronym: ENSAT-HT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Georges Pompidou Hospital (Other); University of Turin, Italy (Other); University of Padova (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: ENSAT-HT-2016-01
Record Dates: First submitted 2016-03-22; First posted 2016-05-13 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: genomics; proteomics; metabolomics; endocrine hypertension; primary aldosteronism; Cushing syndrom; pheochromocytoma
MeSH Terms: conditions — Hypertension; Hyperaldosteronism; Pheochromocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive patients: Diagnostic procedures in patients with hypertension applying omics results
  Interventions: Other: omics

INTERVENTIONS:
Other: omics — diagnostic procedures applying omics results

SUMMARY:
The purpose of this study is to assess the validity and usefulness of omics signatures for improved identification and risk stratification of patients with endocrine hypertension and stratification of patients with primary hypertension.

DETAILED DESCRIPTION:
Arterial hypertension is the most important cause of death in the world. At referral hypertension centers about 25% of patients have a single cause for hypertension, so-called secondary hypertension, mostly of endocrine, adrenal origin (primary aldosteronism, pheochromocytoma/ paraganglioma, Cushing's syndrome). This rate steps up to 50% in patients with drug resistant hypertension. Proper treatment of secondary hypertension improves prognosis considerably but depends on adequate diagnosis. Classically the diagnosis of such forms of hypertension rests on cumbersome biochemical and imaging procedures that may not completely take away uncertainty. Modern '-omics' techniques (genomics, metabolomics, proteomics of plasma and urine) may allow faster and better diagnosis. In addition, they may provide a basis for stratification of hypertensive patients that do not have a identifiable cause of hypertension, so-called primary hypertension. This stratification may help predicting response to antihypertensive drugs and determining prognosis and thus, help to establish personalized medicine in hypertension care.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 75 years old
* A signed and dated informed consent form
* A diagnosis of hypertension defined either as:

  * Use of antihypertensive drug (s)
  * Arterial hypertension: in untreated patients this must be confirmed by daytime ambulatory blood pressure monitoring (ABPM), or home blood pressure monitoring, with blood pressure higher or equal to 135 mmHg for systolic blood pressure and/or higher or equal to 85 mmHg for diastolic blood pressure.

In order to be eligible to participate in the nested case control study, a subject must also meet the following criteria:

- A conformed diagnosis of PA, PPGL or CS for case patients and PHT (exclusion of secondary forms) for their matched counterparts

Exclusion Criteria:

* Any severe comorbid conditions that, according to the attending physician, could decrease the life expectancy to less than 3 years
* Any active malignancy unrelated to adrenal disease or PPGL
* Guardianship for incapacity

A potential control subject who meets any of the following criteria will be excluded from participation in the nested case controlled study in case of:

* Existence of any other forms of secondary hypertension such as renal artery stenosis, renal disease, Munchausen's syndrome in which the patient induces hypertension regardless of method.
* Drug-induced (included factitious use of illicit substances) hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for diagnosis and management of hypertension
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
sensitivities of omics signatures for the diagnosis of subtypes of hypertension | 1 year
  The proportion of patients with various subtypes of endocrine hypertension as identified by omics signature in patients in which subtypes have been identified by usual diagnostic algorithms
specificities of omics signatures for the diagnosis of subtypes of hypertension | 1 year
  The proportion of patients with non-endocrine hypertension as identified by omics signature in patients identified as having non-endocrine hypertension by usual diagnostic algorithms.
positive likelihood ratio | 1 year
  positive likelihood ratios of omics signatures for the diagnosis of subtypes of hypertension
negative likelihood ratio | 1 year
  negative likelihood ratios of omics signatures for the diagnosis of subtypes of hypertension
positive predictive value | 1 year
  positive predictive values of omics signatures for the diagnosis of subtypes of hypertension
negative predictive value | 1 year
  negative predictive values of omics signatures for the diagnosis of subtypes of hypertension

SECONDARY OUTCOMES:
Occurrence of major adverse cardiovascular events (MACE) | within 12 months after baseline
  death, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass grafting (CABG) or need for them, cerebrovascular accident (CVA), hospitalization for acute decompensated heart failure
Left ventricular mass as assessed by echocardiography | 1 year
  Left ventricular mass index measured by ultrasound imaging
Costs | 1 year
  Questionnaires on costs of evaluation, costs of misdiagnosis
Ambulatory blood pressure measurement (ABPM) | 1 year
  ABPM
microalbuminuria | 1 year
  albumin-creatinine ratio in urine
atrial fibrillation | 1 year
  atrial fibrillation as assessed by EKG
RAND-36 | 1 year
  Quality of life assessment by the RAND-36 questionnaire
EQ5D | 1 year
  Quality of life assessment by the EQ5D questionnaire
Hospital Anxiety and Depression Scale (HADS) | 1 year
  Assessment of anxiety and depression by the HADS questionnaire
Cognitive Functioning Questionnaire (CFQ) | 1 year
  Assessment of cognitive functioning by CFQ
Montreal Cognitive Assessment (MOCA) | 1 year
  Assessment of cognitive functioning by MOCA
Home blood pressure measurement (HBPM) | 1 year
  HBPM
number of antihypertensive drugs | 1 year
  number of antihypertensive drugs
defined daily dosages | 1 year
  defined daily dosages of antihypertensive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Maria Christina Zennaro, PhD, Principal Investigator — AP/HECP, Paris
Locations (5):
- European Georges Pompidou Hospital, Paris, France
- Italy (2):
  - University of Padua, Padua
  - University of Torino, Torino
- Raddboudumc, Nijmegen, Gelderland, Netherlands
- University of Glasgow, Glasgow, United Kingdom